CLINICAL TRIAL: NCT04809636
Title: Evaluating the Impact of Incentives on HIV Related Clinical Trial Participation
Brief Title: Evaluating the Impact of Incentives on Clinical Trial Participation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Riverside (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 59270
Record Dates: First submitted 2021-03-02; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Hiv; Aging; Incentives
Keywords: hiv; aging; incentives
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is not an interventional study — While this is not an intervention, there will be separate participants for the survey study and for the other components of the study (focus groups, interviews, conjoint analysis, piloting the vignettes

SUMMARY:
The objective of this study is to investigate the impact of incentives on clinical trial participation. 1) characterize key stakeholders' views on and assessment of incentives, 2) reach consensus among stakeholders on the factors to be considered when choosing incentives and their relative importance, 3) pilot test using vignettes for incentive decision making. We hypothesize that potential study participants make trade-offs regarding the characteristics of a research study when deciding whether to volunteer. This amendment is to document IRB reliance between UCR and USF.

ELIGIBILITY:
Inclusion Criteria:

* people living with HIV
* biomedical HIV researchers
* IRB members/bioethicists involved in HIV research

Exclusion Criteria:

* people under 18 years of age
* people living outside of the United States
* people who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit patient partners, biomedical HIV researchers and IRB members/bioethicists involved in HIV research and patient partners with HIV co-morbidities (depression, heart disease, arthritis). For the patient populations, we will target men (including MSM) and women aging with HIV, cis and transgender women, and youth (age 18+) of color, but participation will be open to everyone over 18 years of age living with HIV who speaks English and live in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
characterize how people living with HIV assess incentives | 3 months
  we will conduct a 20 question quantitative survey of a nationally representative sample of people living with HIV asking about specific study payment information and scenarios
characterize key stakeholders' views on and assessment of incentives | 3 months
  focus groups, and key informant interviews will be used to characterize key stakeholders' (people aging with HIV, IRB members, researchers) views on and assessment of incentives, with qualitative analysis of text done using RaDAR. We will use Conjoint Analysis (CJA) to estimate the relative importance (also called "weight") that participants place on each study characteristic when choosing between different hypothetical studies.
pilot testing vignettes for incentive decision making | 3 months
  We will develop HIV related vignettes (hypothetical scenarios) utilizing the data from outcomes 1 and 2. Specifically, once we have 6 to 8 study characteristics from Aim 2, and the final number of choices (2 - 3) per characteristic, we will use a factorial design to create 25 vignettes (hypothetical scenarios). Individuals from each group (i.e., study participants, researchers, and IRB members) will select the most appropriate incentive from a list of possibilities based on various scenarios. These vignettes will be based on studies identified in the literature and a review of consent forms and created in conjunction with the external advisory board (including pre-testing and revision prior to finalization).

CONTACTS AND LOCATIONS:
Locations (1):
- UC Riverside, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galea JT, Greene KY, Nguyen B, Polonijo AN, Dube K, Taylor J, Christensen C, Zhang Z, Brown B. Evaluating the Impact of Incentives on Clinical Trial Participation: Protocol for a Mixed Methods, Community-Engaged Study. JMIR Res Protoc. 2021 Nov 23;10(11):e33608. doi: 10.2196/33608. PMID 34817381